CLINICAL TRIAL: NCT01073644
Title: Post Marketing Surveillance On The Safety And Tolerability Of Sunitinib Malate (Sutent) For Filipino Patients
Status: Terminated | Type: Observational
Why Stopped: The study was prematurely discontinued due to poor recruitment on 18th April 2013. There were no safety concerns that led to the decision to terminate.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6181118
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-07

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: imatinib resistant or intolerant
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sunitinb malate
  Interventions: Drug: Sunitinib malate

INTERVENTIONS:
Drug: Sunitinib malate — sunitinib 50 mg, 4 weeks on, 2 weeks off
  Other Names: Sutent

SUMMARY:
The primary purpose is to monitor the safety and tolerability and effectiveness of sunitinib malate in the treatment of patients with metastatic renal cell carcinoma and gastrointestinal stromal tumor among filipino patients in usual clinical practice setting.

DETAILED DESCRIPTION:
Open label

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above
* Diagnosed with metastatic renal cell carcinoma or gastrointestinal stromal tumor after imatinib treatment failure or intolerance

Exclusion Criteria:

* Subjects with conditions that are contraindicated with sunitinib malate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be selected by primary care clinic.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2010-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of sunitinib malate as measured by the incidence, severity, seriousness and relatedness to treatment adverse events (AEs), laboratory abnormalities, vital signs (blood pressure) and the use of concomitant medications. | 36 weeks

SECONDARY OUTCOMES:
Effectiveness of sunitinib malate will be measured by the overall response as determined by the objective tumor assessments made according to the Response Evaluation Criteria in Solid Tumors (RECIST). | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Philippines (2):
  - Chong Hua Hospital, Cebu City
  - Private Clinic, Manila

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181118&StudyName=Post%20Marketing%20Surveillance%20On%20The%20Safety%20And%20Tolerability%20Of%20Sunitinib%20Malate%20%28Sutent%29%20For%20Filipino%20Patients%20